CLINICAL TRIAL: NCT02532868
Title: A Phase I Dose Escalation Study of MK0457 Evaluating the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of a 24-Hour Continuous Infusion Given Every 21 Days in Patients With Advanced Cancer
Brief Title: A VX-680 (an Aurora Kinase Inhibitor) Study in Patients With Advanced Cancer (0457-002)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0457-002; 2005_005; NCT00104351 (obsolete NCT alias)
Record Dates: First submitted 2014-07-18; First posted 2015-08-26 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — tozasertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MK-0457 (Experimental): Participants received MK-0457 at assigned dose as a continuous intravenous infusion (CIV) over 24 hours; one group of participants also received MK-0457 100 mg capsules, orally, prior to the CIV.
  Interventions: Drug: MK-0457

INTERVENTIONS:
Drug: MK-0457
  Other Names: VX-680 (an Aurora Kinase Inhibitor)

SUMMARY:
The purpose of this study is to assess the safety and tolerability of MK-0457(VX-680), an Aurora kinase inhibitor, in participants with advanced solid tumors. Bioavailability of the oral formulation will also be assessed. The primary study hypothesis is that administration of MK-0457 is sufficiently safe and tolerated to permit further study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are at least 18 years of age with recurrent or non-responsive solid tumors, or cancers for which standard therapy does not exist.

Exclusion Criteria:

* Patients who have had treatment with any investigational therapy within the past 30 days.
* Patients who have certain types of blood cancers such as leukemia or lymphoma.
* Patients who have uncontrolled congestive heart failure (CHF), chest pains, or had a heart attack within the past 3 months, or have undergone bone marrow or stem cell transplantation.
* Patient is pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2005-05; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants Experiencing Dose-Limiting Toxicities (DLTs) | Up to 21 days

SECONDARY OUTCOMES:
Change in standard uptake value (SUV) in fluorodeoxyglucose positron emission tomography (FDG-PET) scans | Predose, and at end of Cycles 2 and 6 (up to approximately 4 months)
Overall Tumor Response Per Response Evaluation Criteria in Solid Tumors (RECIST) | Pre-dose through post-study visit (up to 3 years)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Traynor AM, Hewitt M, Liu G, Flaherty KT, Clark J, Freedman SJ, Scott BB, Leighton AM, Watson PA, Zhao B, O'Dwyer PJ, Wilding G. Phase I dose escalation study of MK-0457, a novel Aurora kinase inhibitor, in adult patients with advanced solid tumors. Cancer Chemother Pharmacol. 2011 Feb;67(2):305-14. doi: 10.1007/s00280-010-1318-9. Epub 2010 Apr 13. PMID 20386909